CLINICAL TRIAL: NCT05144971
Title: StatStrip A Glucose/Creatinine Meter System Lay User Study Evaluation
Status: Completed | Type: Observational
Sponsor: Nova Biomedical (Industry)
Collaborators: Excellence Medical and Research (Unknown)
Responsible Party: Sponsor
Other Study IDs: NB21-SSA-NA-LAY-FDA
Record Dates: First submitted 2021-11-22; First posted 2021-12-06 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Diabete Mellitus; CKD; ESRD
Keywords: Diabetes; CKD; ESRD; POCT
MeSH Terms: conditions — Diabetes Mellitus; Kidney Failure, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Diagnostic Test: Glucose, Creatinine — Compare diagnostic tests to reference methods

SUMMARY:
The primary objective of this study is to assess the performance of the Nova StatStrip A Glucose/Creatinine Meter System in the hands of the subject (lay user) and compare the result to an accepted Glucose/Creatinine reference method in the hands of a trained technician.

DETAILED DESCRIPTION:
To assess the performance of the StatStrip A Glucose/Creatinine assay in the hands of lay users on capillary whole blood obtained by finger stick and compare with the performance characteristics to a central laboratory traceable reference method.

To assess the Ease of Use of the StatStrip Glucose / Creatinine Meter System in the hands of the intended lay users. Lay users will be provided with all package insert sheets, a Quick Reference Guide and Instructions for Use (IFU) Manual. No training, coaching, or prompting will be provided to the lay users other than clarifying the protocol.

ELIGIBILITY:
Inclusion Criteria:

* Adult subjects (≥ 18 years old) with diabetes.
* Adult subjects (≥ 18 years old) with kidney diseases (CKD, ESRD) and/or in dialysis.
* Adult subjects (≥ 18 years old) that are healthy.
* Subjects willing to complete all study procedures.
* Subjects whose pre-screen glucose or creatinine medical history is deemed of value by the study site
* Subjects able to read, write, speak in English.

Exclusion Criteria:

* Subjects unable to consent to participating in the study.
* Subjects possessing a cognitive disorder or other condition, which, in the opinion of the investigator, would put the person at risk or seriously compromise the integrity of the study.
* Subjects taking prescription anticoagulants (such as Warfarin or Heparin) or has clotting problems that may prolong bleeding.
* Subjects having hemophilia or any other bleeding disorder.
* Subjects having an infection with a blood borne pathogen (e.g. HIV, hepatitis).
* Subjects working for a medical device or diagnostic company.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: A minimum of 150 to a maximum of 200 individual subjects (lay users) will be enrolled.
  Subjects included in the study may be healthy, diabetic or having kidney diseases. The study will be conducted at one study site.
  Adult subjects (≥ 18 years old) of both genders will be included in this study.
  Potential subjects may be screened prior to testing to assess their baseline glucose/creatinine levels. The screening may be done by inspecting medical records.
Sampling Method: Probability Sample
Enrollment: 175 (Actual)
Dates: Start 2021-10-28 (Actual); Primary Completion 2021-12-03 (Actual); Study Completion 2021-12-03 (Actual)

PRIMARY OUTCOMES:
Nova StatStrip A Glucose/Creatinine Meter System | 20 days
  The primary objective of this study is to assess the performance of the Nova StatStrip A Glucose/Creatinine Meter System in the hands of the subject (lay user) and compare the result to an accepted Glucose/Creatinine reference method in the hands of a trained technician.
  The two parameters for the outcome measure in this study are glucose and creatinine. The unit of measure for glucose and creatinine is mg/dL and mmol/L, respectively.

CONTACTS AND LOCATIONS:
Locations (1):
- Excellence Medical Research, Miami Gardens, Florida, United States